CLINICAL TRIAL: NCT05945576
Title: National Cohort on Imprinting Disorders and Their Metabolic Consequences
Brief Title: IDMet (RaDiCo Cohort) (RaDiCo-IDMet)
Acronym: IDMet
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-63
Record Dates: First submitted 2023-06-26; First posted 2023-07-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Silver Russell Syndrome; Beckwith-Wiedemann Syndrome; Transient Neonatal Diabetes Mellitus; Angelman Syndrome; Prader-Willi Syndrome; Temple Syndrome; Kagami-Ogata Syndrome; Pseudohypoparathyroidism; Familial Precocious Puberty
MeSH Terms: conditions — Silver-Russell Syndrome; Beckwith-Wiedemann Syndrome; Angelman Syndrome; Prader-Willi Syndrome; Temple syndrome; Uniparental disomy, paternal, chromosome 14; Pseudohypoparathyroidism; Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Stool collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to describe the natural history of imprinting disorders (IDs) according to their metabolic profile in all patients (adults and children) affected with an ID regardless of the severity of the disease, with a molecular characterization, with a signed informed consent for all subjects, followed in one partner's center.

The main questions it aims to answer are:

* Can we identify common metabolic profiles for all imprinted diseases?
* Which imprinting disorders have an impact on the metabolic profiles of IDs?
* Which are the metabolic risks associated to IDs?
* Can we use the metabolic profiles for the clinical classification and prognosis of IDs?
* Are there common therapeutic approaches for all IDs?

ELIGIBILITY:
Inclusion Criteria:

* Patients (adults and children) affected with an ID regardless of the severity of the disease
* A confirmed diagnosis of ID (based on molecular diagnosis)
* A signed informed consent for adults or signed informed consent of parents/guardians of minors/ protected adult.

Non-Inclusion Criteria:

There are no non-inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (adults and children) affected with an ID regardless of the severity of the disease, with a molecular characterization, with a signed informed consent for all subjects, followed in one partner's center.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The clinical characteristics of IDs in pediatric and adult's patients. | Through study completion, an average of 10 years
The genetic characteristics of IDs in pediatric and adult's patients. | Through study completion, an average of 10 years
The biological characteristics of IDs in pediatric and adult's patients. | Through study completion, an average of 10 years
The morphometric characteristics of IDs in pediatric and adult's patients. | Through study completion, an average of 10 years

SECONDARY OUTCOMES:
Search for an association between the metabolic phenotype of IDs patients' and their biological profil. | At the time of diagnosis (or at first measurement)
Determination of the prevalence of metabolic abnormalities (MA). | At inclusion
Estimation of the risk for metabolic complications such as obesity, diabetes, cardiovascular disease (CVD), metabolic syndrome. | 10 years after
Description of different therapeutic approaches and identification of a common base for all IDs. | Through study completion, an average of 10 years
Variations of quality-of-life scores. | Through study completion, an average of 10 years
Analyse of (epi)genetic mutations transmission in proband and relatives. | Through study completion, an average of 10 years

OTHER OUTCOMES:
Identification of different metabolic profile which allow a clinical classification of IDs. | Through study completion, an average of 10 years
Description and identification of the most relevant biological and clinical practices for diagnostic and follow-up of ID patients. | Through study completion, an average of 10 years
Identification of a group of French patients with the same characteristics. | At inclusion
Search of an association between blood metabolic markers, genetic pattern and gut microbiota. | Through study completion, an average of 10 years
Description of different scientific rational for transferring a therapeutic approach (clinical guidelines) from an ID to another (identification of common phenotype, i.e. metabolic profile). | Through study completion, an average of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Agnès LINGLART, Principal Investigator — Inserm U1169
Locations (18):
- France (18):
  - CHU d'Angers, Angers
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital de la mère et de l'enfant, Limoges
  - Hôpital Femme Mère Enfant, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Brabois, Nancy
  - Hôpital enfant-adolescent, Nantes
  - Hôpital Armand-Trousseau, Paris
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Sud, Rennes
  - Hôpital Civil, Strasbourg
  - Hôpital des Enfants, Toulouse
  - Hôpital Bretonneau, Tours